CLINICAL TRIAL: NCT05310019
Title: Effect of Electroacupuncture on Paresthesias and Functional Changes in Patients Submitted to Bimaxillary Orthognathic Surgery and Mentoplasty
Brief Title: Effect of Electroacupuncture in Patients Submitted Orthognathic Surgery and Mentoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Federal do Ceará (Unknown)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30725720.7.0000.5054.
Record Dates: First submitted 2022-03-02; First posted 2022-04-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Paresthesia; Edema
MeSH Terms: conditions — Paresthesia; Edema | interventions — Physical Therapy Modalities; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy plus Electroacupuncture Group (Experimental): The physiotherapy treatment (50min): warm compress with facial thermal blanket, respiratory muscle mobility training and cervical muscle relaxation, facial lymphatic drainage, start of myolymphokinetic exercises for the orbicularis, zygomatic major and minor muscles, upper lip lifter and nose wing, buccinator and platysma, release of intraoral adhesions, vacuum therapy at 60 mmHg, active exercises free of mandibular movements, maintenance of mandibular opening with wooden tongue depressors. The electroacupuncture treatment lasting another 30 min. Electroacupuncture treatment lasting another 30min. The repetition time of 1 sec; (F1-10 Hz, F2= 45 Hz; 10 mA). Facial acupuncture needles are disposable with 0.20 mm gauge and 10 mm length. Each needle will be inserted at the indicated points, totaling 10 needles and electrodes will be connected to each one. Electrical stimulation will be performed on the face points: E4, Jiachengjiang (extra point), E5, E6, bilaterally and point CV-24.
  Interventions: Other: Physiotherapy and Electroacupuncture
- Physiotherapy Group (Active Comparator): The physiotherapy protocol will be the same as the active group. Protocol: warm compress with facial thermal blanket (5 min), respiratory muscle mobility training and cervical muscle relaxation (5 min) facial lymphatic drainage (10 min), start of myolyphokinetic exercises for the orbicularis oris, zygomatic major and minor, levator labii superioris and nasal ala, buccinator and platysma (5 min), release of intraoral adhesions (5 min) vacuum therapy at 60 mmHg (5 min), active exercises free of mandibular movements of right and left laterality, protrusion and mandibular opening (5 min), maintenance of mandibular opening with wooden tongue depressors (10 min).
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy and Electroacupuncture — TThe physiotherapy treatment (50min): warm compress with facial thermal blanket, respiratory muscle mobility training and cervical muscle relaxation, facial lymphatic drainage, start of myolymphokinetic exercises for the orbicularis, zygomatic major and minor muscles, upper lip lifter and nose wing, buccinator and platysma, release of intraoral adhesions, vacuum therapy at 60 mmHg, active exercises free of mandibular movements, maintenance of mandibular opening with wooden tongue depressors. The electroacupuncture treatment lasting another 30 min. Electroacupuncture treatment lasting another 30min. The repetition time of 1 sec; (F1-10 Hz, F2= 45 Hz; 10 mA). Facial acupuncture needles are disposable with 0.20 mm gauge and 10 mm length. Each needle will be inserted at the indicated points, totaling 10 needles and electrodes will be connected to each one. Electrical stimulation will be performed on the face points: E4, Jiachengjiang (extra point), E5, E6, bilaterally and point CV-24.
  Arms: Physiotherapy plus Electroacupuncture Group
Other: Physiotherapy — The physiotherapy treatment protocol will be divided into 6 meetings: warm compress with facial thermal blanket (5min), respiratory muscle mobility training and cervical muscle relaxation (5min) facial lymphatic drainage (10min), start of myolymphokinetic exercises for the orbicularis oris, zygomatic major and minor muscles, upper lip lifter and nose wing, buccinator and platysma (5 min), release of intraoral adhesions (5min) vacuum therapy at 60 mmHg (5min), active exercises free of mandibular movements (5 min), maintenance of mandibular opening with wooden tongue depressors (10min).
  Arms: Physiotherapy Group

SUMMARY:
Goals. To evaluate the effect of electroacupuncture on paresthesia and myofunctional changes in patients undergoing bimaxillary orthognathic surgery and mentoplasty. Methodology: this is a controlled, randomized, blinded clinical trial. The sample will consist of 62 individuals in each group (general sample = 124 participants). Therefore, 124 young adults, aged between 18 and 50 years, both sexes, with at least 24 teeth, with Class II or III skeletal malocclusion, diagnosed by cephalometric radiographs, who underwent orthognathic surgery in the period from 1 to 30 days before the start of physical therapy, be available to perform the proposed postoperative treatment for six weeks. Participants will be equally and randomly distributed into two experimental groups: GF (Physiotherapy Group), GFE (Physiotherapy plus Electroacupuncture Group). The variables to be studied will be: socioepidemiological data; sensitivity assessment by the Semmes-Weinstein monofilament test; Edema assessment by the MD Anderson Cancer Center Head and Neck Lymphedema protocol, validated in Portuguese; assessment of mandibular movements using a Western-DC digital caliper; Assessment of masticatory function using the Chewing Quality Assessment Questionnaire. Data will be analyzed descriptively and organized into tables. Subsequently, the normality of continuous variables will be tested by the Kolmogorov-Smirnov test. As the variables are normally distributed, we will use parametric tests such as the paired t test, independent t test, ANOVA and Pearson's correlation. Nonparametric tests such as Wilcoxon paired signed rank test, Mann-Whitney U test, Kruskal Wallis test, Spearman correlation test will be used in case of non-normality of continuous variables. The significance level will be adjusted to 5% in all analyses.

DETAILED DESCRIPTION:
Introduction: Among the major oral and maxillofacial surgeries called reconstructive, the one that has become popular in recent years, especially after the mandatory coverage of costs by health plans, was orthognathic surgery, so called because it is a combined procedure between orthodontics and oral and maxillofacial surgery, aiming at the correction of the masticatory system with the objective of reducing the discrepancies related to the jaws and, thus, establishing harmony between the face and the skull. Lesions of the inferior alveolar nerve (INA) are frequent due to its anatomical location, passing through the sagittal osteotomy of the mandibular ramus, where manipulation of the mandibular ramus or the structures that surround the nerve occurs during the operation. Goals. To evaluate the effect of electroacupuncture on paresthesia and myofunctional changes in patients undergoing bimaxillary orthognathic surgery and mentoplasty. Methodology: this is a controlled, randomized, blinded clinical trial. The sample was defined from a pilot study involving ten individuals, considering as an outcome the sensitivity obtained under the same experimental conditions used in this study. A two-way ANOVA with repeated measures considering two factors, group (treatment and control) and irradiation (pre-, post-6 treatment session and post-3 plot) was used to calculate the squared value of the ETA (0.033). The estimated number was 50 individuals per group. For sample calculation, α=0.05 (5% chance of type I error) and 1-β= 0.80 (% of sampling power) were considered. The sample will be increased by 20% to compensate for possible dropouts, resulting in 62 individuals in each group (overall sample = 124 participants). Therefore, 124 young adults, aged between 18 and 50 years, both sexes, with at least 24 teeth, with Class II or III skeletal malocclusion, diagnosed by cephalometric radiographs, who underwent orthognathic surgery in the period from 1 to 30 days before the start of physical therapy, be available to perform the proposed postoperative treatment for six weeks. Participants will be equally and randomly distributed into two experimental groups: GF (Physiotherapy Group), GFE (Physiotherapy plus Electroacupuncture Group). The variables to be studied will be: socioepidemiological data; sensitivity assessment by the Semmes-Weinstein monofilament test; Edema assessment by the MD Anderson Cancer Center Head and Neck Lymphedema protocol, validated in Portuguese; assessment of mandibular movements using a Western-DC digital caliper; Assessment of masticatory function using the Chewing Quality Assessment Questionnaire. Data will be analyzed descriptively and organized into tables. Subsequently, the normality of continuous variables will be tested by the Kolmogorov-Smirnov test. As the variables are normally distributed, we will use parametric tests such as the paired t test, independent t test, ANOVA and Pearson's correlation. Nonparametric tests such as Wilcoxon paired signed rank test, Mann-Whitney U test, Kruskal Wallis test, Spearman correlation test will be used in case of non-normality of continuous variables. The significance level will be adjusted to 5% in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing bimaxillary orthognathic surgery and mentoplasty;
* Aged between 18 and 50 years;
* Both of genders,
* Having at least 24 teeth, with Class II or III skeletal malocclusion;
* Diagnosed by cephalometric radiographs, who have performed the surgery in the period from 1 to 45 days before the beginning of physiotherapy;
* Be available to perform the proposed postoperative treatment at the Clinic School of Physiotherapy of the Estácio do Ceará University Center for six weeks;
* Agree to participate in the research;
* Sign the term of free and clear clarification.

Exclusion Criteria:

* Individuals with cleft lip or palate, previous orthopedic and/or rheumatologic diseases that may have repercussions on the face such as facial fractures, facial palsy, systemic lupus erythematosus, neurological alteration due to injury or compression of the facial or trigeminal nerve;
* Patients with chronic lymphedema, individuals treated or undergoing cancer treatment, syndromic, with local vascular changes or who have undergone previous surgeries on the face such as bichectomy, TMJ surgery, with the exception of tooth extraction without associated nervous impairment, who performed other surgical procedures combined with orthognathic;
* Patients who use botulinum toxin for the treatment of temporomandibular dysfunction and esthetics;
* Patients who presented postoperative complications such as infectious processes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
sensitivity assessment | the sensitivity assessment at 6 months
  Using the Semmes-Weinstein monofilament test

SECONDARY OUTCOMES:
measure range of motion | The range of motion at at 6 months
  range of motion (measure with digital calipers)
measure edema | the edema assessment at 6 months
  The edema will be measured with the aid of a measuring tape.
measure functionality | measure Functionality at 6 months
  The functionality will be measured with Chewing Quality Assessment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Itana L Spinato, Principal Investigator — Universidade Federal do Ceará
Locations (1):
- Clinic School of the University Center Estácio do Ceará, Fortaleza, Ceará, Brazil